CLINICAL TRIAL: NCT02504853
Title: Natural History and Genetics of Food Allergy and Related Conditions
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150162; 15-I-0162
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2025-12-09 (Actual); Status verified 2025-12-04

CONDITIONS: Food Allergy; Loeys-Dietz Syndrome; Atopic Dermatitis; Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; Loeys-Dietz Syndrome; Atopic Dermatitis; TGFbeta; Natural History
MeSH Terms: conditions — Food Hypersensitivity; Loeys-Dietz Syndrome; Dermatitis, Atopic; Eosinophilic Esophagitis; Camurati-Engelmann Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Affected Genetic: Have a suspected genetic or congenital disorder potentially associated with food allergy or related condition, as determined by the principal investigator (PI) or associate investigators (AIs).
- Affected Non-Syndromic Food: Individuals with a clinical history of immediate hypersensitivity reaction to foods and sensitized to food allergen(s) as evidenced by SPT or allergen-specific IgE testing.
- Allergic GI Disease: Individuals with a diagnosis or clinical suspicion of eosinophilic esophagitis (EoE), as determined by the principal investigator (PI) or associate investigators (AIs).
- Unaffected Relative / Healthy Volunteer: Unaffected relatives are relatives of affected; unaffected by food allergy or the genetic condition under study. Healthy volunteers are not related to affected and serve as controls.

SUMMARY:
Background:

- About 15 million Americans have a food allergy. Because there are no cures or effective prevention or treatment for food allergies, researchers want to learn more about them.

Objective:

- To learn more about the causes and effects of food allergy and related conditions.

Eligibility:

* People ages 2 99 who have food allergy and/or a related genetic or other condition
* Their relatives
* Healthy relatives and volunteers

Design:

* Participants will have at least 3 visits over 1 2 years, and then once a year for up to 12 years. Each may last a day or longer.
* Participants will be screened with medical history, physical exam, and questionnaires.
* Participants may have the following:
* Blood tests
* Allergy skin prick tests: Drops of allergens are placed on the back or arm. The skin is scratched under each drop.
* Leukapheresis: blood is taken from a needle in one arm, passed through a machine, and returned through a needle in the other arm.
* X-rays
* Esophageal string test: One end of a string is taped to the cheek and the other end is packed into a capsule. When the capsule is swallowed, the string unwinds; it is left in for at least 1 hour.
* EGD and colonoscopy: Biopsies are taken from the gastrointestinal system.
* Tiny biopsies of skin
* Photographs of the body
* Collection of cells through:
* Swab of nose, inside of cheek, or skin
* Gentle skin scrape
* Tape stripping: piece of tape is put on the skin and pulled off.

DETAILED DESCRIPTION:
There are approximately 15 million Americans, including 6 million children, who have a potentially life-threatening food allergy. The prevalence of this disease has increased over the last three decades, in both the United States and other developed countries. There are no cures or effective prevention or treatment strategies for food allergy. Moreover, little is known about the factors that account for the rising prevalence and severity of these diseases in recent years. Both genetic and environmental factors likely contribute to the development of food allergy, but the complex interaction between these variables has frustrated efforts to elucidate pathogenesis and develop mechanism-targeted therapies. Children with food allergy are 2 to 4 times more likely to be diagnosed with asthma or other allergic conditions than children without food allergy, and food allergy may also be an important trigger for atopic dermatitis and eosinophilic esophagitis. The Laboratory of Allergic Diseases within the National Institute of Allergy and Infectious Diseases has a longstanding interest in the genetics and pathogenesis of allergic inflammatory disorders, and with the National Institutes of Health Clinical Center, it provides the ideal environment for the proposed translational studies. In this study, we will: (1) investigate the key genetic, cellular, immunologic, and biochemical pathways that lead to the development of food allergy, and (2) identify biomarkers that predict the clinical course and natural history of patients with food allergy.

Subjects eligible for enrollment in this study include children and adults with food allergy and patients with a known/suspected genetic or congenital disorder potentially associated with these phenotypes. Unaffected relatives (children and adults) of an enrolled subject and healthy volunteers (children and adults) will also be eligible for enrollment as controls. Most participants will be followed for 2 years, although participants with an identified genetic or congenital disorder and a subset of participants with food allergy may be followed until this study ends (up to 25 years).

Data obtained from analysis of blood, skin, saliva, stool, gastrointestinal biopsies, and other specimens will be used to explore the immunologic, biochemical, microbial, and genetic basis of food allergy. Results of research studies will be correlated with the scope and severity of their clinical phenotype, their response to treatment, and the natural history of their allergic disease(s).

ELIGIBILITY:
* GENERAL INCLUSION CRITERIA:

All participants must meet the following criteria:

1. Be 2 to 99 years-old at the time of enrollment for participants who will be seen at the NIH CC; be 0 (newborn) to 99 years-old at the time of enrollment for participants who will submit mail-in samples or participate in telehealth visits. Only viable neonates will be enrolled.
2. Willing to allow storage of blood, buccal swabs, saliva, nasal swabs, stool samples, and other clinically appropriate tissue specimens for future use in medical research
3. Required to have a primary care or other physician who will manage all health conditions related or unrelated to the study objectives

ADDITIONAL INCLUSION CRITERIA FOR AFFECTED PARTICIPANTS

In addition to the general criteria listed above, affected participants must meet 1 of the following criteria:

1. Have a clinical history of an immediate hypersensitivity reaction to food(s) and be sensitized to food allergen(s) (as evidenced by positive SPT or allergen-specific IgE testing)
2. Be sensitized (as evidenced by positive SPT or allergen-specific IgE testing) to food allergen(s) but have no overt clinical history of IgE-mediated symptoms when they eat that food(s)
3. Have a suspected genetic or congenital disorder potentially associated with food allergy or related condition, as determined by the principal investigator (PI) or associate investigators (AIs)
4. Have a diagnosis of eosinophilic esophagitis (EoE), or clinical suspicion for EoE as determined by the principal investigator (PI) or associate investigators (AIs)
5. Have a history of atopic dermatitis based on self-report or physician assessment.

ADDITIONAL INCLUSION CRITERIA FOR UNAFFECTED RELATIVES:

In addition to the general criteria listed above, unaffected relatives must meet the following criteria:

1. Be a relative of an affected participant
2. Be unaffected by food allergy (as determined by clinical history and/or allergy testing) or be unaffected by the genetic condition under study

ADDITIONAL INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS

In addition to the general criteria listed above , healthy volunteers must meet the following criteria:

1. Be unrelated to an affected participant
2. Be unaffected by food allergy (as determined by clinical history and/or allergy testing) or be unaffected by the genetic condition under study

ADDITIONAL PROCEDURE- SPECIFIC INCLUSION CRITERIA:

The following additional inclusion criteria apply for participants undergoing leukapheresis:

1. Age greater than or equal to 18 years
2. Stable hematologic parameters (definition: white blood cell count > 2,500/microL, hemoglobin > 10 g/dL, and platelet count > 75,000/microL)

GENERAL EXCLUSION CRITERIA:

Participants will be excluded for any of the following:

* Presence of conditions that, in the judgment of the investigator or the referring physician, may put the participant at undue risk or make them unsuitable for participation in the study.
* Inability to participate for the duration of the study.
* The PI deems that participation in the study would not be expected to advance the study goals.

ADDITIONAL PROCEDURE- SPECIFIC EXCLUSION CRITERIA

Additional exclusion criteria apply for unaffected relatives and healthy volunteers who are undergoing endoscopy with biopsies for research purposes. Unaffected relatives and healthy volunteers will be excluded from participating in this procedure if they meet any of the following criteria:

1. uncontrolled asthma or Grade 3 or higher by the American Society of Anesthesiologist s. Physical Status Classification System (http://www.asahq.org/resources/clinicalinformation/.asa-physical-status-classification-system)
2. history of adverse reaction to conscious sedation or general anesthesia required for endoscopy
3. hemoglobin < 11 g/dL
4. platelet count < 100,000 microL
5. PT INR >1.3 or PTT prolonged by > 3 seconds
6. pregnant or breastfeeding
7. viral screens positive for HIV or hepatitis B or C
8. severe unstable myocardial ischemia or cardiomyopathy
9. severe hypoxemia due to chronic pulmonary disease
10. recent abdominal surgery
11. anticoagulant therapy that cannot be interrupted
12. history of reflux disease within the last 3 years or use of acid-suppression medication (including over-the-counter medications such as Tums, Rolaids, Zantac, Prilosec OTC, or Prevacid OTC) within the last 2 months
13. chronic GI or immunologic disease
14. clinically indicated EGD or colonoscopy within the past 12 months
15. use of systemic or inhaled corticosteroids within the past 4 months
16. have a history of EGID including EoE
17. younger than 18 years of age

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2015-07-29 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Investigate the key genetic, cellular, immunologic, microbial, and biochemical pathways that lead to the development of food allergy | 06/15/2025
  Investigate the key genetic, cellular, immunologic, microbial, and biochemical pathways that lead to the development of food allergy
Identify biomarkers that predict the clinical course and natural history of patients with food allergy | 06/15/2025
  Identify biomarkers that predict the clinical course and natural history of patients with food allergy

SECONDARY OUTCOMES:
The prevalence of eosinophilic GI disease in patients who might be considered to be at high risk for these conditions, including those patients with atopic dermatitis and/or multiple food sensitivities/allergies | 06/15/2025
In vitro testing of novel therapies for food allergy using cells and other biological specimens obtained from patients with food allergy | 06/15/2025
Identification of nutritional deficiencies and their effect on the growth and overall health of patients with food allergy and related conditions | 06/15/2025

CONTACTS AND LOCATIONS:
Overall Officials: Pamela A Guerrerio, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months after publication.
Access Criteria: Data that requires public reporting to be deposited in public databases, data required to be in publications, and data required for collaborations.

REFERENCES:
- [Background] Boyce JA, Assa'ad A, Burks AW, Jones SM, Sampson HA, Wood RA, Plaut M, Cooper SF, Fenton MJ, Arshad SH, Bahna SL, Beck LA, Byrd-Bredbenner C, Camargo CA Jr, Eichenfield L, Furuta GT, Hanifin JM, Jones C, Kraft M, Levy BD, Lieberman P, Luccioli S, McCall KM, Schneider LC, Simon RA, Simons FE, Teach SJ, Yawn BP, Schwaninger JM. Guidelines for the diagnosis and management of food allergy in the United States: summary of the NIAID-sponsored expert panel report. Nutr Res. 2011 Jan;31(1):61-75. doi: 10.1016/j.nutres.2011.01.001. No abstract available. PMID 21310308
- [Background] Noval Rivas M, Burton OT, Wise P, Zhang YQ, Hobson SA, Garcia Lloret M, Chehoud C, Kuczynski J, DeSantis T, Warrington J, Hyde ER, Petrosino JF, Gerber GK, Bry L, Oettgen HC, Mazmanian SK, Chatila TA. A microbiota signature associated with experimental food allergy promotes allergic sensitization and anaphylaxis. J Allergy Clin Immunol. 2013 Jan;131(1):201-12. doi: 10.1016/j.jaci.2012.10.026. Epub 2012 Nov 30. PMID 23201093
- [Background] Frischmeyer-Guerrerio PA, Guerrerio AL, Oswald G, Chichester K, Myers L, Halushka MK, Oliva-Hemker M, Wood RA, Dietz HC. TGFbeta receptor mutations impose a strong predisposition for human allergic disease. Sci Transl Med. 2013 Jul 24;5(195):195ra94. doi: 10.1126/scitranslmed.3006448. PMID 23884466
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-I-0162.html